CLINICAL TRIAL: NCT03195569
Title: To Predict Efficacy by Detecting Circulating Endothelial Cell Subsets and Blood Perfusion Parameters Changes in Vivo Tumor in Study of QL1101 and Avastin® in Patients With Non-squamous Non-small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Collaborators: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: QL1101
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Non Small Cell Lung Cancer
Keywords: QL1101 Avastin® Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Experimental group: QL1101 + paclitaxel/carboplatin:subjects are given 15 mg/kg QL1101 on Day 1 of each cycle with every 3 weeks as a cycle, respectively combined with paclitaxel/carboplatin for 6 cycles.
  Interventions: Drug: QL1101; Drug: Paclitaxel; Drug: Carboplatin
- Control group: Avastin® + paclitaxel/carboplatin:subjects are given 15 mg/kg Avastin® on Day 1 of each cycle with every 3 weeks as a cycle, respectively combined with paclitaxel/carboplatin for 6 cycles.
  Interventions: Drug: Avastin®; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: QL1101 — targeted vascular endothelial growth factor (VEGF) monoclonal antibodies
  Groups: Experimental group
Drug: Avastin® — targeted vascular endothelial growth factor (VEGF) monoclonal antibodies
  Other Names: bevacizumab
  Groups: Control group
Drug: Paclitaxel — 175 mg/m2, IV following investigational product on day 1 of each 21 day cycle.
Drug: Carboplatin — AUC 5 IV, following paclitaxel on day 1 of each 21 day cycle.

SUMMARY:
To reveal changes of peripheral markers and blood perfusion parameters in vivo tumor in the study of QL1101 and Avastin® in patients with Non-squamous Non-small Cell Lung Cancer

DETAILED DESCRIPTION:
The study is QL1101-002 additional research, by detecting the blood circulating endothelial cells and blood perfusion parameters change within tumors early prediction efficacy and drug resistance.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years and ≤75 years;
* Patients with histologically or cytologically confirmed inoperable locally advanced (Stage IIIb, not suitable for multidisciplinary treatment), metastatic (Stage IV), or relapsed non-squamous cell non-small cell lung cancer. Diagnostic result of non-squamous cell non-small cell lung cancer obtained based on sputum cytology should be immunohistochemically confirmed. If a variety of tumor ingredients are mixed, the main cell types should be classified;
* ECOG score of 0-1 points;
* At least one measurable lesion can be evaluated according to RECIST1.1 criteria;
* Patients who have not received systemic anti-tumor therapy of locally advanced or metastatic non-squamous non-small cell lung cancer (if the subject received adjuvant therapy after completing the radical treatment of early non-small cell lung cancer, but then the disease relapsed, the subject can be enrolled. In this case, the end time of the adjuvant therapy is required to be more than 6 months from the time of the first administration of this study, and various toxic reactions resulting from the adjuvant therapy should have recovered (≤ Grade 1 by CTCAE 4.03 criteria, except for alopecia);
* Expected survival time ≥24 weeks;

Exclusion Criteria:

* Central squamous cell carcinoma, and mixed gland squamous cell carcinoma with squamous cell as the main ingredient;
* ALK fusion gene is known to be positive;
* Medical history or examination shows thrombotic disease within 6 months prior to screening;
* Imaging shows signs of tumor invasion of large vessels, and the investigator or radiologist must exclude patients whose tumor has been completely close to or surrounded or invaded the lumen of large vessels (e.g., the superior pulmonary artery or superior vena cava);
* Patients with a past history of symptomatic brain metastases or meningeal metastases, or spinal cord compression;
* Patients who received palliative radiotherapy for bone lesions outside the chest within 2 weeks prior to the first dose of the study drug;
* Patients who received major surgical procedures (including thoracotomy), or suffered from major trauma (such as fractures) within 28 days
* prior to screening, or need to undergo major surgery during the expected study treatment period;
* Patients who received a minor surgical procedure within 48 hours prior to the first treatment with Anivitis® QL1101 (the investigator judges whether there is bleeding tendency);

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with Non-squamous Non-small Cell Lung Cancer,who should meet the eligibility criteria.Because the study is QL1101-002 additional research, all people meet QL1101-002 clinical research requirements
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-06-12 (Estimated); Study Completion 2018-12-10 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 18 weeks
  The actual endpoint is best response seen during the study
Number of circulating endothelial cell subsets | different time points before and after one week of treatment of QL1101 or avastin, an expected average of 2 weeks
  To detect the number of circulating activated endothelial cell (aCECs) by flow cytometry

SECONDARY OUTCOMES:
The strength of intratumoral blood perfusion index(BV,BF,PS and MTT) | different time points before and after 3 weeks of treatment QL1101 or avastin, an expected average of 6 weeks
  To detect the strength of intratumoral blood perfusion index(BV,BF,PS and MTT) by CT perfusion imaging
Disease control rate | 3 months, 6 months, 9 months, 1 year
  DOR is defined as the time from the first tumor evaluation as CR or PR to the first evaluation as PD or death
Treatment-emergent adverse events | 18 week
  Assessment following therapy with either QL1101 or avastin

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tainjin, China